CLINICAL TRIAL: NCT03423017
Title: Brainstem Dysfunction Involvement in the Pathogenesis of Pierre Robin Sequence
Acronym: DYSROBIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0816
Record Dates: First submitted 2018-01-12; First posted 2018-02-06 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Pierre Robin Sequence; Brainstem Dysfunction
Keywords: Pierre Robin sequence; Brainstem; pathogenesis; swallowing; apnea
MeSH Terms: conditions — Pierre Robin Syndrome; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pierre Robin sequence (Other): Infants with PRS : retrognathism, glossoptosis, cleft palate
  Group 1a : isolated PRS Group 1b : PRS with bone disease or collagen disease (Stickler) Group 1c : syndromic PRS or associated PRS without bone disease or collagen disease
  Interventions: Other: Recording of data
- Superior airway obstruction, AWO (Other): Infants with AWO : laryngomalacia, tracheal stenosis, laryngeal stenosis, others etiology
  Interventions: Other: Recording of data
- Healthy infants (Other): Healthy infants : siblings of sudden unexpected death of the infant
  Interventions: Other: Recording of data

INTERVENTIONS:
Other: Recording of data — Recording during one hospitalization of 48 hours between birth and 2 months of life and one hospitalization of 24 hours between 6 and 10 months of life
  * General data: age, term of birth, birth weight, gender, diseases, weight and size at recording, cranial perimeter, food, drugs : first and second visit
  * Respiratory rate, respiratory signs, stridor : first and second visit
  * 24h holter-ECG : first and second visit
  * 24h impedance pH-metry : first visit
  * Nocturne polysomnography : 50% prone position, 50% supine : sleep analyze, obstructive apnea hypopnea index (OAHI), central apnea index (CAI), periodical breathing, micro arousals index, non-nutritive swallowing analyze,(mental region electromyogram) : first and second visit
  * 24 h gaz exchanges : mean, maximal PtcCO2 and % of time spent above 50 mmHg , SpO2 under 90%, 85% et 80% and desaturations index : first and second visit
  * succimetry procedure : at first visit only between birth and 2 months
  Arms: Pierre Robin sequence; Superior airway obstruction, AWO
Other: Recording of data — Recording during one hospitalization of 48 hours between birth and 2 months of life
  * General data: age, term of birth, birth weight, gender, diseases, weight and size at recording, cranial perimeter, food, drugs
  * Respiratory rate, respiratory signs, stridor
  * 24h holter-ECG
  * 24h impedance pH-metry
  * Nocturne polysomnography : 100% supine position : sleep analyze, obstructive apnea hypopnea index (OAHI), central apnea index (CAI), periodical breathing, micro arousals index, non-nutritive swallowing analyze,(mental region electromyogram)
  * 24 h gas exchanges : mean, maximal PtcCO2 and % of time spent above 50 mmHg , SpO2 under 90%, 85% et 80% and desaturations index
  * Succimetry procedure : at first visit only between birth and 2 months
  Arms: Healthy infants

SUMMARY:
Introduction Pierre Robin Sequence, PRS, incidence is about one hundred births per year in France. The main neonatal clinical manifestations are secondary to airway obstruction and food difficulties related to swallowing disorders. Despite recent progress, the pathogenesis of PRS is not fully understood.

The hypothesis is that brainstem dysfunction, BSD, plays a central role in the pathogenesis of PRS.

The purpose of the study is to achieve a complete evaluation of BSD to specify its role in the pathogenesis of PRS.

The primary objective is to compare central apnea index (CAI) of infants with PRS with those of infants with isolated airway obstruction (AWO) and those of healthy infants in order to clarify the direct role of BSD.

Material and Methods This prospective interventional study will be carried out in Lyon at the Hôpital Femme-Mère-Enfant and in Paris at the Hôpital Necker-Enfants Malades for 2 years. 3 groups of patients will be studied: PRS, 50 patients, AWO, 50 patients and healthy, 30 patients, included before 2 months of life. Infants will be followed for a maximum of 10 months. The evaluations will be carried out for 48 hours between birth and 2 months of life and then for 24 hours between 6 and 10 months of life for PRS and AWO group. Concerning the healthy group, the evaluation will be carried out during 48h during a single hospitalization before 2 months. Polysomnography, holter-ECG, 24h gas exchange, impedance-pH monitoring and mental region EEG will be performed. The central apnea index (mean number per hour), obstructive apnea index, non-nutritive swallowing index (NNS), gastroesophageal reflux and NNS-respiration coordination will be assessed for each stage of sleep and compared between the three groups of patients.

ELIGIBILITY:
Inclusion Criteria for the group 1

- infants with PRS

Inclusion Criteria for the group 2 - infant with isolated airway obstruction

Inclusion Criteria for the group 3

- healthy infant : siblings of sudden unexpected death of the infant or with any known pathology

Inclusion Criteria for the 3 groups

* During one hospitalization or program for one hospitalization
* Parental consent
* Social safety affiliation

Exclusion Criteria:

* Birth before 37 SA
* Neonatal complication
* Group 2 only: AWO with neurological disease including brainstem dysfunction
* Group 3 only : AWO, ENT disease or syndromic disease, neurological disease including brainstem dysfunction, Intra uterine growth retardation

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Central apnea index (CAI) (mean number per hour) | 2 months of life during one nocturne polysomnography
  To compare central apnea index (CAI) (mean number per hour), according to the ASSM guidelines 2007, recording by one nocturne polysomnography, between 3 groups of infants by sleep step, between birth and 2 months of life, in order to clarify the direct role of BSD.
  According to the ASSM guidelines 2007, the central apnea index is measured : mean number of central apnea per hour.

SECONDARY OUTCOMES:
Obstructive apnea hypopnea index (OAHI)(mean number per hour) | 2 months
  To compare obstructive apnea hypopnea index (OAHI)(mean number per hour) according to the guidelines ASSM 2007, recording by one nocturne polysomnography, between 3 groups of infants by sleep step, between birth and 2 months of life According to the ASSM guidelines 2007, the obstructive apnea hypopnea index is measured: mean number of obstructive apnea and hypopnea per hour.
Comparison of OAHI(mean number per hour) and CAI | between 6 and 10 months of life
  To compare obstructive apnea hypopnea index (OAHI)(mean number per hour) and central apnea index (CAI) (mean number per hour), between PRS group and AWO group by sleep step between 6 and 10 months of life
  According to the ASSM guidelines 2007, the obstructive apnea hypopnea index, mean number of obstructive apnea and hypopnea per hour, and the central apnea index are measured, mean number of central apnea per hour.
Micro arousals index (mean number per hour) | up to 2 months of life
  To compare micro arousals index (mean number per hour) between the 3 groups by sleep step between birth and 2 months of life and between PRS group and AWO group between 6 and 10 months of life to clarify the role of BSD in sleep microstructure
  According to the ASSM guidelines 2007, micro arousals index (mean number per hour) are measured.
Micro arousals index (mean number per hour) | up to 10 months of life
  To compare micro arousals index (mean number per hour) between the 3 groups by sleep step between birth and 2 months of life and between PRS group and AWO group between 6 and 10 months of life to clarify the role of BSD in sleep microstructure
  According to the ASSM guidelines 2007, micro arousals index (mean number per hour) are measured.
Non-nutritive swallowing index (NNS) and apnea secondary to non-nutritive swallowing | up to 2 months of life
  To compare non-nutritive swallowing index (NNS) and apnea secondary to non-nutritive swallowing between the 3 groups by sleep step between birth and 2 months of life and between PRS group and AWO group between 6 and 10 months of life to clarify the role of BSD in swallowing disorders and NNS-respiration coordination
  non-nutritive swallowing index (NNS), mean number per hour, and apnea secondary to non-nutritive swallowing, mean number per hour, monitoring by the mental region EEG and the one nocturne polysomnography
Non-nutritive swallowing index (NNS) and apnea secondary to non-nutritive swallowing | up to 10 months of life
  To compare non-nutritive swallowing index (NNS) and apnea secondary to non-nutritive swallowing between the 3 groups by sleep step between birth and 2 months of life and between PRS group and AWO group between 6 and 10 months of life to clarify the role of BSD in swallowing disorders and NNS-respiration coordination
  non-nutritive swallowing index (NNS), mean number per hour, and apnea secondary to non-nutritive swallowing, mean number per hour, monitoring by the mental region EEG and the one nocturne polysomnography
Positive and negative pressures, their temporal organizations evaluated using succimetry procedure between the 3 groups of patients at 0 and 2 months of life | up to 2 months of life
  Compare the positive and negative pressures, their temporal organizations evaluated using succimetry procedure between the 3 groups of patients at 0 and 2 months of life.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Femme Mère Enfant, Bron
  - APHP-Necker, Paris

IPD SHARING:
Plan to Share IPD: Undecided